CLINICAL TRIAL: NCT00001439
Title: A Phase I Study of gp100 Human Melanoma Peptide Vaccine With Incomplete Freund's Adjuvant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 950145; 95-C-0145
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-05

CONDITIONS: Melanoma
Keywords: Cancer; Immunotherapy
MeSH Terms: conditions — Melanoma; Neoplasms | interventions — PMEL protein, human

INTERVENTIONS:
Biological: gp100 human melanoma peptide

SUMMARY:
This is a phase I study of melanoma tumor antigen peptide vaccines. The nine amino acid peptides representing HLA-A2 restricted T cell epitope of the melanoma antigen, gp100 will be administered to patients emulsified in Incomplete Freund's Adjuvant, (IFA). The study is designed to evaluate the toxicity, immunologic effects and potential therapeutic role of repeated doses of gp100 peptide vaccines administered subcutaneously.

Immune reactivity to the gp100 epitope peptides will be monitored in all patients by analysis of melanoma-specific T cell precursor frequency prior to and after immunization.

DETAILED DESCRIPTION:
This is a phase I study of melanoma tumor antigen peptide vaccines. The nine amino acid peptides representing HLA-A2 restricted T cell epitope of the melanoma antigen, gp100 will be administered to patients emulsified in Incomplete Freund's Adjuvant, (IFA). The study is designed to evaluate the toxicity, immunologic effects and potential therapeutic role of repeated doses of gp100 peptide vaccines administered subcutaneously.

Immune reactivity to the gp100 epitope peptides will be monitored in all patients by analysis of melanoma-specific T cell precursor frequency prior to and after immunization.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Metastatic melanoma that is HLA-A2 positive.

No primary melanoma of ocular or mucosal origin.

Measurable or resected metastatic disease required.

PRIOR/CONCURRENT THERAPY:

BIOLOGIC THERAPY: No prior (greater than 30 days) or concurrent Biologic Therapy.

CHEMOTHERAPY: No prior (greater than 30 days) or concurrent chemotherapy.

ENDOCRINE THERAPY: No prior (greater than 30 days) or concurrent hormone therapy.

No requirement for steroids.

RADIOTHERAPY: No prior (greater than 30 days) or concurrent radiotherapy.

SURGERY: Not specified.

PATIENT CHARACTERISTICS:

Age: 18 and over.

Performance Status: ECOG 0 or 1.

Life Expectancy: More than 3 months.

HEMATOPOIETIC: No coagulation disorder.

HEPATIC:

Bilirubin no greater than 2.0 mg/dL.

No Hepatitis BsAg antibody.

RENAL: Creatinine no greater than 2.0 mg/dL.

CARDIOVASCULAR: No major cardiovascular illness.

PULMONARY: No major respiratory illness.

OTHER:

No previous allergic reaction to incomplete Freund's adjuvant.

HIV negative.

No active systemic infection.

Not pregnant or lactating.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 255
Dates: Start 1995-06; Study Completion 2000-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Rosenberg SA. Cancer vaccines based on the identification of genes encoding cancer regression antigens. Immunol Today. 1997 Apr;18(4):175-82. doi: 10.1016/s0167-5699(97)84664-6. No abstract available. PMID 9136454
- [Background] Rosenberg SA. Development of cancer immunotherapies based on identification of the genes encoding cancer regression antigens. J Natl Cancer Inst. 1996 Nov 20;88(22):1635-44. doi: 10.1093/jnci/88.22.1635. PMID 8931607
- [Background] Rosenberg SA, Yang JC, Schwartzentruber DJ, Hwu P, Marincola FM, Topalian SL, Restifo NP, Dudley ME, Schwarz SL, Spiess PJ, Wunderlich JR, Parkhurst MR, Kawakami Y, Seipp CA, Einhorn JH, White DE. Immunologic and therapeutic evaluation of a synthetic peptide vaccine for the treatment of patients with metastatic melanoma. Nat Med. 1998 Mar;4(3):321-7. doi: 10.1038/nm0398-321. PMID 9500606